CLINICAL TRIAL: NCT00109837
Title: A Phase II Study of Double Induction Chemotherapy for Newly Diagnosed Non-L3 Adult Acute Lymphoblastic Leukemia With Investigation of Minimal Residual Disease and Risk of Relapse Following Maintenance Chemotherapy
Brief Title: S0333 Combination Chemotherapy in Treating Patients With Newly Diagnosed Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S0333; U10CA032102 (NIH); S0333 (Other: SWOG)
Record Dates: First submitted 2005-05-03; First posted 2005-05-04 (Estimated); Results first posted 2012-08-23 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Leukemia
Keywords: L1 adult acute lymphoblastic leukemia; L2 adult acute lymphoblastic leukemia; untreated adult acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Filgrastim; Cyclophosphamide; Cytarabine; Daunorubicin; Dexamethasone; Doxorubicin; Leucovorin; Mercaptopurine; Methotrexate; Mitoxantrone; Asparaginase; Prednisone; Thioguanine; Vincristine; Radiotherapy; Allopurinol; Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Induc x2, Consol, Maint (Experimental): Induc 1: Allopurinol; Daunorubicin; Vincristine; Prednisone; asparaginase; Bactrim Induc 2: Allopurinol; cytarabine; Dexamethasone; filgrastim; mitoxantrone; Methotrexate; leucovorin Consol: Cyclophosphamide; cytarabine; 6-mercaptopurine; Methotrexate; filgrastim Maint:Course 1: 6-mercaptopurine; Methotrexate Course 2: Vincristine; doxorubicin; Dexamethasone Course 3: Cyclophosphamidee; thioguanine; cytarabine Course 4: 6-mercaptopurine; methotrexate
  Interventions: Biological: filgrastim; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin; Drug: dexamethasone; Drug: doxorubicin; Drug: leucovorin; Drug: mercaptopurine; Drug: methotrexate; Drug: mitoxantrone; Drug: Asparaginase; Drug: prednisone; Drug: thioguanine; Drug: vincristine; Radiation: radiation therapy; Drug: allopurinol; Drug: bactrim

INTERVENTIONS:
Biological: filgrastim — As needed per physician discretion
Drug: cyclophosphamide — Cyclophosphamide Consolidation: 650 mg/m2; IV; days 1, 15, 29 Post-consolidation course 3: 650 mg/m2; IV; day 1
Drug: cytarabine — Induction 2: 3 g/m2; IV over 3 hrs; days 1-5 Consolidation: 75 mg/m2/d; IV push; days 2-5 and 16-19 Post-consolidation course 3: 75 mg/m2/d; IV push; days 3-6 and 10-13
Drug: daunorubicin — Induction: 60 mg/m2/d; IV; days 1, 2, and 3
Drug: dexamethasone — Induction 2: 0.1% QID; eye drops; days 1-6 Post consolidation course 2: 10 mg/m2/d; PO; days 1-28
Drug: doxorubicin — Post consolidation: 25 mg/m2; IV; days 1, 8, 15, and 22
Drug: leucovorin — For CNS during induction: 5 mg every 6 hrs for 4 doses; PO; days 1, 4, 8, 11, etx.; after methotrexate if WBC < 3,000
Drug: mercaptopurine — Consolidation: 60 mg/m2; PO; days 1-28 Post-consolidation course 1: 60 mg/m2/d; PO; days 1-63 Post-consolidation course 4: 60 mg/m2/d; PO; daily for 2 yrs
Drug: methotrexate — Consolidation: 12 mg; intrathecal or intraventricularly; days 2, 9, 16, and 23 Post-consolidation course 1: 20 mg/m2/wk; PO; days 1, 8 15, 22, 29, 36, 43, 50, 57 Post-consolidation course 4: 20 mg/m2; PO; weekly for 2 yrs
Drug: mitoxantrone — Induction 2: 80 mg/m2; IV; day 3
Drug: Asparaginase — Induction: 2,000 IU/m2; IM or IV; day 15
Drug: prednisone — Induction: 60 mg/m2/d; PO or IV; days 1-35
Drug: thioguanine — Post-consolidation course 3: 60 mg/m2/d; PO; days 1-14
Drug: vincristine — Induction: 1.4 mg/m2/d (2 mg max); IV; days 1, 8, 15, 22
Radiation: radiation therapy — For CNS during consolidation: cranial radiation after blasts are no longer present in spinal fluid. Total dose of 1800 cGy over 2 wks in 10 fractions of 180 cGy 5 days/wk.
Drug: allopurinol — 300 mg/d PO Days 1-7
Drug: bactrim — 1 double strenth tablet 2x/d, 2x/wk, PO, begin with prednisone

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy), and giving the drugs in different combinations may kill more cancer cells.

PURPOSE: This phase II trial is studying how well combination chemotherapy works in treating patients with newly diagnosed acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the probability of 1-year continuous complete remission in patients with newly diagnosed acute lymphoblastic leukemia treated with first induction chemotherapy comprising daunorubicin, vincristine, prednisone, and pegaspargase; and second induction chemotherapy comprising high-dose cytarabine and mitoxantrone.

Secondary

* Determine the frequency and severity of toxic effects of these induction regimens followed by consolidation therapy comprising cyclophosphamide, cytarabine, mercaptopurine, and methotrexate and maintenance chemotherapy comprising mercaptopurine, methotrexate, vincristine, doxorubicin, dexamethasone, cyclophosphamide, thioguanine, and cytarabine in these patients.

Other objectives (if funding allows):

* To evaluate in a preliminary manner the significance of detecting minimal residual disease as a prognostic factor for survival and relapse-free survival of patients receiving chemotherapy
* To evaluate in a preliminary manner the pattern of gene expression of patients entered onto the trial and its relationship to cytogenetics/FISH risk classification, overall survival, and relapse-free survival

OUTLINE: This is a multicenter study.

* First induction chemotherapy: Patients receive daunorubicin IV on days 1-3; vincristine IV on days 1, 8, 15, and 22; prednisone IV or orally on days 1-28, followed by a taper to day 35; and pegaspargase IV or subcutaneously (SC) on day 15. Patients with CNS leukemia also receive methotrexate intrathecally (IT) or intraventricularly twice weekly and oral leucovorin calcium four times daily for 4 doses after each administration of methotrexate. When blasts are no longer present in the spinal fluid, patients receive methotrexate IT or intraventricularly once weekly for 4 weeks and then once monthly for 1 year.

Patients are reevaluated on day 28. Patients who achieve A1 bone marrow status and B1 peripheral blood status or those with resistant disease proceed to second induction therapy.

* Second induction chemotherapy: Patients receive high-dose cytarabine IV on days 1-5; mitoxantrone IV on day 3; and filgrastim (G-CSF) SC or IV beginning on day 7 and continuing until blood counts recover. Patients with CNS leukemia also receive methotrexate and leucovorin calcium as in first induction chemotherapy.

Patients are reevaluated on day 28. Patients who achieve A1 bone marrow status and B1 peripheral blood status with no extramedullary disease (other than CNS involvement) proceed to consolidation chemotherapy. Patients with resistant disease OR Philadelphia chromosome- or BCR/ABL-positive disease are removed from the study after receiving double induction chemotherapy.

* Consolidation chemotherapy: Patients receive cyclophosphamide IV on days 1, 15, and 29; cytarabine IV on days 2-5 and 16-19; oral mercaptopurine on days 1-28; and methotrexate IT or intraventricularly on days 2, 9, 16, and 23. Patients with CNS leukemia also undergo cranial radiotherapy once daily, 5 days a week, for 2 weeks.

Patients in complete remission proceed to maintenance chemotherapy.

* Maintenance chemotherapy:

  * Course 1: Patients receive oral mercaptopurine on days 1-63 and oral methotrexate on days 1, 8, 15, 22, 29, 36, 43, 50, and 57. Patients proceed to course 2 after blood counts recover.
  * Course 2: Patients receive vincristine IV and doxorubicin IV on days 1, 8, 15, and 22 and oral dexamethasone on days 1-28. Patients proceed to course 3 after blood counts recover.
  * Course 3: Patients receive cyclophosphamide IV on day 1; oral thioguanine on days 1-14; and cytarabine IV on days 3-6 and 10-13. Patients proceed to course 4 after blood counts recover.
  * Course 4: Patients receive oral mercaptopurine once daily for 2 years and oral methotrexate once weekly for 2 years.

Treatment continues in the absence of disease relapse or unacceptable toxicity.

After completion of study therapy, patients are followed every 3 months for 1 year, every 6 months for 1 year, and then annually for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Morphologically confirmed acute lymphoblastic leukemia (ALL), meeting any of the following criteria:

  * FAB class L1 or L2 disease
  * Mixed lineage ALL
* Ph-negative/BCR/ABL-negative
* Newly diagnosed disease
* Patients with the following diagnoses are not eligible:

  * FAB class L3 ALL
  * Non-Hodgkin's lymphoma
  * Chronic myelogenous leukemia in lymphoid blast crisis
  * Mixed lineage acute myeloid leukemia
  * Acute minimally differentiated myeloid leukemia (M0)
* Must be registered on protocols SWOG-9007 AND SWOG-S9910

PATIENT CHARACTERISTICS:

Age

* 18 to 64

Performance status

* Zubrod 0-3

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* No chronic liver disease
* Hepatitis panel, including hepatitis B and C, negative

  * History of hepatitis A with positive antibody allowed

Renal

* Creatinine ≤ 1.5 times upper limit of normal OR
* Creatinine clearance > 60 mL/min

Cardiovascular

* Left ventricular function normal

  * Ejection fraction ≥ 50% by MUGA or 2-dimensional echocardiogram
* No symptomatic congestive heart failure
* No coronary artery disease
* No cardiomyopathy
* No uncontrolled arrhythmia

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* HIV negative
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer in complete remission

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior remission induction chemotherapy for ALL

  * Prior hydroxyurea to control WBC count allowed

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No other prior treatment for ALL

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2005-04; Primary Completion 2010-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Radich, MD, Study Chair — Fred Hutchinson Cancer Center; Frederick R. Appelbaum, MD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (78):
- United States (78):
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Shawnee Mission Medical Center, Shawnee Mission, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Independence Regional Health Center, Independence, Missouri
  - Truman Medical Center - Hospital Hill, Kansas City, Missouri
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - St. Joseph Medical Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Parvin Radiation Oncology, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Frontier Cancer Center, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - AnMed Cancer Center, Anderson, South Carolina
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Treatment included:
  Induc 1: Allo; Dauno; Vin; Pred; asparag; Bactrim Induc 2: Allo; AraC; Dex; GCSF; Mitx; Meth; leuc; Meth Consol: cyclo; AraC; 6-mercapto; Meth; GCSF Maint:Course 1: 6-mercapto; Meth 20 Course 2: Vincristine; Adriamycin; Dex Course 3: Cyclo; 6-thio; AraC Course 4: 6-mercapto; meth
Period: Overall Study
Arm/Group | Treatment
Started | 79
Eligible | 78
Eligible and Ph- | 61
Eligible and Ph- and Treated | 60
Completed | 56
Not Completed | 23
Not completed — Adverse Event | 2
Not completed — Refusal unrelated to adverse effects | 1
Not completed — Death | 1
Not completed — BCR/ABL+ or Ph+ | 17
Not completed — Not treated | 1
Not completed — Ineligible | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 60
Age, Continuous [Median (Full Range); unit: years] | 42 [18 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 40
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Continuous Complete Remission at 1 Year
Description: A patient has a continuous complete remission at 1 year if they achieve a CR and are alive 365 days after registering to the study.
Time Frame: After induction, after consolidation, every 3 months during maintenance, and every three months after off treatment for up to a year
Population: Eligible, Ph-, treated, and evaluable patients
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 58
participants | 21
Statistical Analysis 1: Comparison: Treatment; The regimen would be of no further interest if the true 1-year continuous complete remission (CCR) rate was less than 45% (null). Sample size was chosen for an alternative of 65%, power of 92% and type-1 error of 4.6%; Test type: Superiority or Other; Proportion in 1-year CCR = 0.36, 95% CI 1-sided [lower limit 0.25], Standard Deviation 0.06

2. Secondary Outcome: Toxicity
Description: Number of patients with Grade 3-5 adverse events that are related to study drug by given type of adverse event
Time Frame: Patients were assessed for adverse events after the induction cycle
Population: Eligible patients who started therapy
Measure: Number; unit: Participants with a given type of AE
Groups:
- Induction: One induction cycle with allopurinol, daunorubicin, vincristine, prednisone, amd PEG- L-asparaginase.
Arm/Group | Induction
Number analyzed (Participants) | 74
Participants with a given type of AE
  ALT, SGPT (serum glutamic pyruvic transaminase) | 17
  AST, SGOT (serum glut oxaloacetic transaminase) | 13
  Albumin, serum-low (hypoalbuminemia) | 3
  Alkaline phosphatase | 2
  Anorexia | 2
  Ascites (non-malignant) | 1
  Bilirubin (hyperbilirubinemia) | 6
  Calcium, serum-low (hypocalcemia) | 7
  Cholecystitis | 1
  Cholesterol, serum-high (hypercholesterolemia) | 2
  Coagulation-Other (Specify) | 1
  Colitis, infectious (e.g., Clostridium difficile) | 1
  Constipation | 1
  DIC (disseminated intravascular coagulation) | 2
  Death not assoc with CTCAE term-Multi-organ fail | 1
  Edema: limb | 1
  Fatigue (asthenia, lethargy, malaise) | 3
  Febrile neutropenia | 18
  Fever (in the abs of neutropenia) | 1
  Fibrinogen | 11
  Glucose, serum-high (hyperglycemia) | 16
  Glucose, serum-low (hypoglycemia) | 1
  Hemoglobin | 33
  Hypertension | 2
  Hypotension | 3
  Hypoxia | 2
  Ileus, GI (functional obstruction of bowel) | 1
  Infec(doc clin or mibio) w/ Gr 3/4 neut-Anal | 1
  Infec(doc clin or mibio) w/ Gr 3/4 neut-Bladder | 1
  Infec(doc clin or mibio) w/ Gr 3/4 neut-Blood | 11
  Infec(doc clin or mibio) w/ Gr 3/4 neut-Bronchus | 1
  IInfec(doc clin or mibio) w/ Gr 3/4 neut-Catheter | 1
  Infec(doc clin or mibio) w/ Gr 3/4 neut-Eye NOS | 1
  Infec(doc clin or mibio) w/ Gr 3/4 neut-Lung | 1
  Infec(doc clin or mibio) w/ Gr 3/4 neut-Nose | 1
  Infec(doc clin or mibio) w/ Gr 3/4 neut-Pharynx | 1
  Infec(doc clin or mibio) w/ Gr 3/4 neut-Ur tract | 2
  Infec with nor ANC or Gr 1/2 neut-Lung (pneumonia) | 2
  Infection-Other (Specify) | 1
  Leukocytes (total WBC) | 43
  Lipase | 1
  Liver dysfunction/failure (clinical) | 2
  Lymphopenia | 19
  Magnesium, serum-high (hypermagnesemia) | 1
  Mucositis/stomatitis (clinical exam) - Oral cavity | 2
  Mucositis/stomatitis (funct/symp) - Oral cavity | 1
  Mucositis/stomatitis (func/symp) - Pharynx | 1
  Muscle weak,gen spec area-Whole body | 2
  Nausea | 3
  Neuropathy: motor | 1
  Neutrophils/granulocytes (ANC/AGC) | 47
  Pain - Abdomen NOS | 1
  Pain - Bone | 1
  Pain - Neck | 1
  Pancreatic endocrine: glucose intolerance | 1
  Pancreatitis | 1
  Phosphate, serum-low (hypophosphatemia) | 1
  Platelets | 44
  Potassium, serum-high (hyperkalemia) | 1
  Potassium, serum-low (hypokalemia) | 7
  Rash/desquamation | 1
  Renal failure | 2
  Sodium, serum-low (hyponatremia) | 6
  Thrombosis/thrombus/embolism | 1
  Thrombotic microangiopathy | 2
  Triglyceride, serum-high (hypertriglyceridemia) | 1
  Tumor lysis syndrome | 5
  Typhlitis (cecal inflammation) | 1
  Uric acid, serum-high (hyperuricemia) | 1
  Vomiting | 1

ADVERSE EVENTS:
Time Frame: While the patient is on treatment until resolution of acute toxicities with maximum grade reported
Description: Regular investigator assessments are reported after each cycle of protocol treatment
Groups:
- First Induction: One induction cycle with allopurinol, daunorubicin, vincristine, prednisone, amd PEG- L-asparaginase.
- Second Induction: A second induction cycle with allopurinol , dexamergasone, G-CSF, high-dose ara-C and mitoxantrone
- Consolidation: Patients who had a CR after induction could receive one course of consolidation therapy consisting of cyclophosphamide, ara-C, 6-mercaptopurine, G-CSF and methotrexate
- Maintenance: Patient with a CR after consolidation could receive up to four courses of maintenance. Course 1 included 6-mercaptopurine and methotrexate. course 2 included vincristine, adriamycin, and dexamethasone. course 3 included cyclophosphamide, 6-thioguanine, and ara-C. course 4 included 6-mercaptopurine and methotrexate
Arm/Group | First Induction | Second Induction | Consolidation | Maintenance
Serious Adverse Events (participants affected / at risk) | 2/75 | 2/56 | 1/33 | 0/12
Other Adverse Events (participants affected / at risk) | 71/75 | 54/56 | 33/33 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | First Induction (N=75) | Second Induction (N=56) | Consolidation (N=33) | Maintenance (N=12)
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Death not associated with CTCAE term - Multi-organ failure (General disorders) | 1 | 0 | 0 | 0
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Blood (Infections and infestations) | 0 | 1 | 0 | 0
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Lung (pneumon (Infections and infestations) | 0 | 1 | 0 | 0
Hemorrhage/bleeding associated with surgery, intra-operative or post-operative (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Leukocytes (total WBC) (Investigations) | 0 | 0 | 1 | 0
Platelets (Investigations) | 0 | 0 | 1 | 0
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | First Induction (N=75) | Second Induction (N=56) | Consolidation (N=33) | Maintenance (N=12)
Febrile neutropenia (Blood and lymphatic system disorders) | 19 | 30 | 2 | 0
Hemoglobin (Blood and lymphatic system disorders) | 43 | 35 | 21 | 6
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1
Supraventricular and nodal arrhythmia - Sinus tachycardia (Cardiac disorders) | 4 | 5 | 0 | 0
Constipation (Gastrointestinal disorders) | 27 | 6 | 3 | 3
Diarrhea (Gastrointestinal disorders) | 18 | 23 | 2 | 3
Distention/bloating, abdominal (Gastrointestinal disorders) | 5 | 0 | 0 | 0
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal-Other (Specify) (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Heartburn/dyspepsia (Gastrointestinal disorders) | 6 | 0 | 2 | 0
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 6 | 8 | 0 | 1
Mucositis/stomatitis (functional/symptomatic) - Oral cavity (Gastrointestinal disorders) | 5 | 4 | 0 | 1
Nausea (Gastrointestinal disorders) | 31 | 26 | 14 | 4
Pain - Abdomen NOS (Gastrointestinal disorders) | 6 | 6 | 0 | 2
Pain - Oral cavity (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 15 | 19 | 7 | 3
Edema: limb (General disorders) | 11 | 7 | 0 | 0
Fatigue (asthenia, lethargy, malaise) (General disorders) | 37 | 36 | 19 | 7
Fever (in the absence of neutropenia, where neutropenia is defined as ANC lt1.0 x 10e9/L) (General disorders) | 4 | 12 | 4 | 3
Pain - Pain NOS (General disorders) | 0 | 0 | 0 | 1
Pain-Other (Specify) (General disorders) | 0 | 0 | 0 | 2
Rigors/chills (General disorders) | 11 | 22 | 0 | 0
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 4 | 0 | 0 | 0
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 0 | 3 | 0 | 1
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Blood (Infections and infestations) | 11 | 11 | 0 | 0
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Lung (pneumon (Infections and infestations) | 0 | 0 | 0 | 1
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Skin (celluli (Infections and infestations) | 0 | 0 | 0 | 1
Infection with unknown ANC - Mucosa (Infections and infestations) | 0 | 0 | 0 | 1
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 38 | 27 | 9 | 3
AST, SGOT (serum glutamic oxaloacetic transaminase) (Investigations) | 37 | 22 | 8 | 3
Alkaline phosphatase (Investigations) | 21 | 9 | 0 | 3
Amylase (Investigations) | 4 | 0 | 0 | 0
Bilirubin (hyperbilirubinemia) (Investigations) | 28 | 15 | 5 | 1
CPK (creatine phosphokinase) (Investigations) | 0 | 0 | 0 | 1
Creatinine (Investigations) | 8 | 5 | 2 | 0
Fibrinogen (Investigations) | 14 | 0 | 0 | 0
Leukocytes (total WBC) (Investigations) | 43 | 34 | 21 | 9
Lymphopenia (Investigations) | 20 | 15 | 9 | 3
Metabolic/Laboratory-Other (Specify) (Investigations) | 5 | 0 | 0 | 1
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 49 | 39 | 28 | 8
PTT (Partial thromboplastin time) (Investigations) | 5 | 0 | 0 | 0
Platelets (Investigations) | 48 | 43 | 24 | 7
Weight loss (Investigations) | 10 | 8 | 0 | 1
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 18 | 23 | 8 | 2
Anorexia (Metabolism and nutrition disorders) | 11 | 14 | 5 | 2
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 29 | 20 | 4 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 30 | 16 | 5 | 2
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 4 | 0 | 2 | 0
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 5 | 0 | 0 | 0
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 0 | 6 | 3 | 0
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 0 | 3 | 0 | 0
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 6 | 0 | 0 | 0
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 19 | 14 | 6 | 2
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 16 | 13 | 3 | 0
Tumor lysis syndrome (Metabolism and nutrition disorders) | 5 | 0 | 0 | 0
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 4 | 0 | 0 | 0
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscle weakness, generalized or specific area (not due to neuropathy) - Whole body/generalized (Musculoskeletal and connective tissue disorders) | 9 | 3 | 4 | 0
Pain - Back (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0 | 0
Pain - Bone (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 1
Pain - Joint (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0 | 0
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0 | 1
Dizziness (Nervous system disorders) | 8 | 6 | 2 | 2
Neuropathy: motor (Nervous system disorders) | 4 | 0 | 2 | 1
Neuropathy: sensory (Nervous system disorders) | 24 | 15 | 4 | 5
Pain - Head/headache (Nervous system disorders) | 13 | 14 | 8 | 4
Taste alteration (dysgeusia) (Nervous system disorders) | 0 | 4 | 0 | 2
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 14 | 4 | 0 | 2
Mood alteration - anxiety (Psychiatric disorders) | 5 | 0 | 0 | 1
Mood alteration - depression (Psychiatric disorders) | 0 | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 2 | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 6 | 7 | 3 | 2
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 0 | 0
Mucositis/stomatitis (clinical exam) - Pharynx (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 0 | 0
Mucositis/stomatitis (functional/symptomatic) - Pharynx (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 28 | 17 | 4 | 3
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Skin and subcutaneous tissue disorders) | 0 | 3 | 4 | 0
Pruritus/itching (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 5 | 11 | 0 | 2
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 0 | 5 | 0 | 0
Hemorrhage/Bleeding-Other (Specify) (Vascular disorders) | 0 | 3 | 0 | 0
Hypertension (Vascular disorders) | 5 | 0 | 0 | 1
Hypotension (Vascular disorders) | 5 | 11 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No